CLINICAL TRIAL: NCT06403293
Title: Influence of Sonic Activation of Epoxy Resin and Calcium Silicate Sealer on Post-Operative Pain: A Patient-Blinded, Randomised Clinical Trial
Brief Title: Influence of Sonic Activation of Root Sealers on Post-Operative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Merve Sari, Assistant Professor, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 280424
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Post Operative Pain; Apical Periodontitis
Keywords: apical periodontitis; post operative pain; calcium silicate; endoactivator
MeSH Terms: conditions — Pain, Postoperative; Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patients were blinded to the chosen root canal sealer and activation protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AH Plus-NA (Experimental): AH Plus was mixed according to the manufacturer's instructions. The R40 gutta-percha (VDW) was coated with the sealer and inserted into the canal, and the root canals were filled using the single cone technique (SCT). The sealer was not activated.
  Interventions: Procedure: Root canal treatment (AH Plus-NA)
- AH Plus- EA (Experimental): An EA 25/04 tip was coated with AH Plus and activated in the root canals for 10 seconds. Then, the R40 gutta-percha was coated with the sealer and inserted into the canal, and the root canals were filled using SCT.
  Interventions: Procedure: Root canal treatment (AH Plus-EA)
- BC-NA (Experimental): The ready-to-use EndoSequence BC was injected into the root canals and no activation was performed. Then, the R40 gutta-percha was inserted into the canali and the root canals were filled using SCT.
  Interventions: Procedure: Root canal treatment (BC-NA)
- BC-EA (Experimental): EndoSequence BC was injected into the root canals. An EA 25/04 tip was inserted 2 mm beyond the WL and activated for 10 s. Then, the R40 gutta-percha was inserted into the canal and the root canals were filled using SCT.
  Interventions: Procedure: Root canal treatment (BC-EA)

INTERVENTIONS:
Procedure: Root canal treatment (AH Plus-NA) — Root canal treatment procedures explained in arm descriptions.
  Arms: AH Plus-NA
Procedure: Root canal treatment (AH Plus-EA) — Root canal treatment procedures explained in arm descriptions.
  Arms: AH Plus- EA
Procedure: Root canal treatment (BC-NA) — Root canal treatment procedures explained in arm descriptions.
  Arms: BC-NA
Procedure: Root canal treatment (BC-EA) — Root canal treatment procedures explained in arm descriptions.
  Arms: BC-EA

SUMMARY:
Aim: This clinical study aims to compare post-operative pain after single-visit root canal treatment of teeth with asymptomatic apical periodontitis using epoxy-resin based AH Plus and calcium silicate based Endosequence BC sealers with or without sonic activation.

Materials and Methods: The study included 72 individuals having one first or second mandibular premolar tooth with asymptomatic apical periodontitis. They were randomly divided into 4 groups according to the root canal sealer (AH Plus or Endosequence BC) and activation protocol (sonic activation or non-activation) (n=18). Participants were ask to rate their post-operative pain intensity on a NRS scale as none, minimal, moderate, or severe after 24 h, 48 h, 72 h and 7 days following treatment. Patients were also asked to record the number of prescribed analgesic medication tablets (ibuprofen 400 mg) taken. The collected data were statistically analyzed at 0.05 significance level.

DETAILED DESCRIPTION:
Root Canal Treatment After inferior alveolar nervus block anesthesia with 4% Articaine with 1:100,000 adrenaline, the tooth was isolated with a rubber dam. The access cavity was opened using high-speed diamond round burs under water cooling. The working length (WL) was set at 0.5 mm shorter than the 0.0 reading using a 15 K-type file and apex locator (Morita Root ZX, Japan) and checked with radiographs. The root canals were prepared with Resiproc (Resiproc, VDW, Munich, Germany) R25 and R40 files, respectively, at the WL using the crown down technique. A total of 20 mL of 2.5% sodium hypochlorite (NaOCl) was used with a 30-gauge needle (Max-i-Probe; Dentsply Sirona) during preparation. 5 mL of distilled water was left in the canal for 1 min to neutralize the effect of NaOCl, and then the root canals were irrigated with 3 ml of 17% ethylene diamine tetra acetic acid (EDTA). EDTA was activated for 3 × 20s with the EA 25/04 tip 2 mm shorter than the WL. The EA tip was used with 2-4 mm vertical strokes. The root canals were irrigated with 5 mL distilled water and dried with paper points.

The subjects were divided into four groups for root filling. Randomization was performed using online software (www.randomizer.org) with a four-block-sized block randomization technique to ensure even distribution between the groups (allocation ratio 1:1:1:1). A co-investigator managed the allocation and reported the allocated treatment procedure to the operator. The operator could not be blinded due to the different stages of the treatment protocols. The patients were blinded to the chosen root canal sealer and activation protocol.

ELIGIBILITY:
Inclusion Criteria:

* Mandibular first and second premolar teeth diagnosed with asymptomatic apical periodontitis
* Single rooted teeth with a single canal.

Exclusion Criteria:

* Previous root canal treatment
* Use of any analgesic or antibiotics in the last 7 days
* Symptomatic teeth
* Sinus tract
* Presence of advanced periodontal problem (probing depth >4 mm)
* Complications during treatment such as broken file, ledging
* Teeth with extensive coronal destruction.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
post operative pain | 1 week
  All participants were given a questionnaire based on a 0-10 numeric rating scale (NRS), with 0 indicating no pain and 10 indicating the worst pain. Patients recorded their pain on days 1, 2, 3 and 7 after treatment. Pain intensity was rated into 4 categories using the NRS. None: (NRS 0); Mild (NRS 1-3); Moderate (NRS 4-7); Severe (NRS 8-10).

CONTACTS AND LOCATIONS:
Locations (1):
- Mustafa Kemal University, Hatay, Antakya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fonseca B, Coelho MS, Bueno CEDS, Fontana CE, Martin AS, Rocha DGP. Assessment of Extrusion and Postoperative Pain of a Bioceramic and Resin-Based Root Canal Sealer. Eur J Dent. 2019 Jul;13(3):343-348. doi: 10.1055/s-0039-3399457. Epub 2019 Dec 3. PMID 31794999
- [Result] Gundogar M, Sezgin GP, Kaplan SS, Ozyurek H, Uslu G, Ozyurek T. Postoperative pain after different irrigation activation techniques: a randomized, clinical trial. Odontology. 2021 Apr;109(2):385-392. doi: 10.1007/s10266-020-00553-5. Epub 2020 Sep 11. PMID 32915346
- [Result] Aslan T, Donmez Ozkan H. The effect of two calcium silicate-based and one epoxy resin-based root canal sealer on postoperative pain: a randomized controlled trial. Int Endod J. 2021 Feb;54(2):190-197. doi: 10.1111/iej.13411. Epub 2020 Oct 17. PMID 32929721
- [Result] Graunaite I, Skucaite N, Lodiene G, Agentiene I, Machiulskiene V. Effect of Resin-based and Bioceramic Root Canal Sealers on Postoperative Pain: A Split-mouth Randomized Controlled Trial. J Endod. 2018 May;44(5):689-693. doi: 10.1016/j.joen.2018.02.010. Epub 2018 Mar 20. PMID 29571915
- [Result] Wiesse PEB, Silva-Sousa YT, Pereira RD, Estrela C, Domingues LM, Pecora JD, Sousa-Neto MD. Effect of ultrasonic and sonic activation of root canal sealers on the push-out bond strength and interfacial adaptation to root canal dentine. Int Endod J. 2018 Jan;51(1):102-111. doi: 10.1111/iej.12794. Epub 2017 Jun 19. PMID 28543092
- [Result] Lopes FC, Zangirolami C, Mazzi-Chaves JF, Silva-Sousa AC, Crozeta BM, Silva-Sousa YTC, Sousa-Neto MD. Effect of sonic and ultrasonic activation on physicochemical properties of root canal sealers. J Appl Oral Sci. 2019 Sep 9;27:e20180556. doi: 10.1590/1678-7757-2018-0556. PMID 31508791
- [Derived] Yilmaz K, Sari M. Influence of sonic activation of epoxy-resin and calcium silicate sealer on postoperative pain: a patient-blinded, parallel group, randomized clinical trial. BMC Oral Health. 2024 Oct 23;24(1):1268. doi: 10.1186/s12903-024-05049-0. PMID 39443924